CLINICAL TRIAL: NCT03851926
Title: Hypofractionated Radiotherapy for Prostate Cancer in 20 Sessions
Brief Title: Hypofractionated Radiotherapy for Prostate Cancer
Acronym: HRT20
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Nicolas Feltes, Principal Investigator, Consorci Sanitari de Terrassa
Other Study IDs: ONCORTCST2019-1
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: HYPOFRACTIONED
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Hypofractionated volumetric radiotherapy in 20 fractions — Hypofractionated radiotherapy at 3 Gy per fraction for localized prostate cancer.

SUMMARY:
Radiotherapy is a standard definitive treatment for men with localized prostate cancer.

Recent improvements in technology allow high doses of radiation to be delivered to the prostate in less days with lower doses to surrounding healthy tissues, trying to reduce side effects.

This study is being proposed to evaluate the use of moderate hypofractionated volumetric radiotherapy in localized prostate cancer patients and assessing treatment -related later adverse events using the CTCAE 4.0

DETAILED DESCRIPTION:
Recent evidence suggests that the same or better outcomes might be achieved in prostate cancer by ussing a higher dose of radiation per fraction ( 3Gy) with the consequent decrease in total days Quality of life outcomes as well as gastrointestinal and genitourinary late toxicities will be analyzed.

It is thought that this regimen will produce comparable findings and would result in substantial health care cost savings, as well as, be more convenient for patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of adenocarcinoma of the prostate by biopsy
* Performance Status 0-2
* Signed informed consent form

Exclusion Criteria:

* Positive lymph-nodes or metastatic disease from prostate cancer on imaging studies
* Anticoagulant treatment, individual assessment of antiplatelet therapy
* Previous pelvic radiotherapy
* Previous surgery for prostate cancer
* Previous transurethral resection of the prostate
* History of Crohn's Disease or Ulcerative Colitis
* Antecedents of rectal fistulas in the last 10 years
* Previous significant urinary obstructive symptoms
* Previous chemotherapeutic treatments
* Non-compliance with constraints established in this protocol (see special section

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events assessed by CTCAE v4.0 | Participants should be followed continuously, for the duration of 10 years
  Number of patients with treatment-related adverse events as assessed by Common Toxicity Criteria for Adverse Effects v4.0

SECONDARY OUTCOMES:
Biochemical relapse free survival | Participants should be followed continuously, for the duration of 10 years
  By Phoenix definition ( Nadir + 2 ng/ml) Participants should be followed at baseline and follow-up, for the duration of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: NICOLAS FELTES, Study Director — Consorci Sanitari de Terrassa
Locations (1):
- Hospital de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided